CLINICAL TRIAL: NCT00132418
Title: Double-blind, Randomized, Placebo-controlled Study of Enbrel (Etanercept) in the Treatment of Rheumatoid Arthritis Subjects With Comorbid Disorders
Brief Title: Study of Enbrel in Rheumatoid Arthritis (RA) Subjects With Comorbid Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20021629
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis and at least 1 qualifying comorbid condition (diabetes, chronic pulmonary disease, recent infection); RA; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Diabetes Mellitus | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- Enbrel (Experimental): Enbrel
  Interventions: Drug: Enbrel

INTERVENTIONS:
Drug: Enbrel — Enbrel
  Arms: Enbrel
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of this study was to evaluate the safety of Enbrel (etanercept) in rheumatoid arthritis (RA) subjects with greater than or equal to 1 documented comorbid disease (diabetes mellitus; chronic pulmonary disease; pneumonia within the last year; or recurrent bronchitis, sinusitis, or urinary tract infection) that might increase infection risk.

ELIGIBILITY:
Inclusion Criteria: - Active RA - Documented comorbid condition (diabetes mellitus requiring insulin or oral hypoglycemic agents; chronic pulmonary disease; history of pneumonia in the last year; or recurrent bronchitis, sinusitis or urinary tract infection) - Able to self-inject study drug Exclusion Criteria: - Previous use of anti-tumor necrosis factor (TNF) monoclonal antibody - Receipt of anti-CD4 or diphtheria interleukin-2 fusion protein within the previous 6 months with subsequent abnormal absolute T cell count - Receipt of intra-articular corticosteroids within 2 weeks before screening - Receipt of cyclosporine, thalidomide or azathioprine within 4 weeks before screening - Significant concurrent medical diseases (serious infection; open cutaneous ulcers; current antibiotic treatment; myocardial infarction [MI] within 12 months of screening; angina pectoris; uncontrolled hypertension; cancer; or HIV positive)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2000-04; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Incidence of medically important infections, defined as infections that result in hospitalization or treatment with intravenous antibiotics | 16 weeks

SECONDARY OUTCOMES:
Infections associated with antimicrobial use; physical examination, vital signs, clinical laboratory assessments; symptom assessment, withdrawals, deaths, and serious adverse events | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Weisman MH, Paulus HE, Burch FX, Kivitz AJ, Fierer J, Dunn M, Kerr DR, Tsuji W, Baumgartner SW. A placebo-controlled, randomized, double-blinded study evaluating the safety of etanercept in patients with rheumatoid arthritis and concomitant comorbid diseases. Rheumatology (Oxford). 2007 Jul;46(7):1122-5. doi: 10.1093/rheumatology/kem033. Epub 2007 Apr 29. PMID 17470434
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20021629.pdf
- See also: FDA-approved Drug Labeling — http://www.enbrel.com/